CLINICAL TRIAL: NCT04950595
Title: Defining the Satiety Characteristics of Plant-based Mince in Comparison to Standard Beef Mince: Does Plant-based Mince Make You Feel Fuller for Longer?
Brief Title: Plant-based Mince vs Beef Mince: Does One Make You Feel Fuller for Longer?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government)
Collaborators: v2food (https://www.v2food.com/) (Unknown)
Responsible Party: Principal Investigator, Bradley Klingner, Research Technician, Commonwealth Scientific and Industrial Research Organisation, Australia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: VTF001
Record Dates: First submitted 2021-06-10; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: Single-centre, single-blinded, randomised, cross-over trial.
Who Masked: Participant
Masking Description: Single (participants are blinded). The provision of the two test meals will be randomised and participants will be blinded to which meal they will receive (although we acknowledge they may be able to distinguish them by taste).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beef mince group (Experimental): The test meal provided at lunch will be made up of 45% beef mince, with all remaining ingredients the same as the other arm.
  Interventions: Other: Beef mince
- Plant-based mince group (Experimental): The test meal provided at lunch will be made up of 45% plant-based mince, with all remaining ingredients the same as the other arm.
  Interventions: Other: Plant-based mince

INTERVENTIONS:
Other: Plant-based mince — Spaghetti bolognaise meal made with plant-based mince
  Arms: Plant-based mince group
Other: Beef mince — Spaghetti bolognaise meal made with beef mince
  Arms: Beef mince group

SUMMARY:
This project will provide preliminary evidence to support whether V2 plant-based mince could contribute to increased satiety following a meal, which may assist in a weight reduction dietary regime when substituted for standard beef mince.

DETAILED DESCRIPTION:
Growing concerns about the sustainability and environmental impacts of red meat consumption have resulted in the increased uptake of plant-based red meat substitutes by consumers worldwide. In addition to the environmental benefits of these products, it has also been argued that they have the potential to offer additional health benefits. One such health benefit, and the focus of this study, is the potential for plant-based meats to produce a greater satiating effect in comparison to traditional meat products, and therefore potentially assist in supporting weight loss or weight maintenance in the longer term.

To address this question, the investigators will assess the effect of substituting V2 mince for beef mince in a standard pasta meal on both the amount of the meal consumed and on feelings of fullness in the period after eating, as assessed by both subjective reporting, objective (biochemical) measures and the amount consumed at a subsequent meal occasion. The results of this study will provide proof-of-concept evidence of the potential enhanced satiating effects of V2 mince, and therefore whether it could potentially assist in a weight reduction dietary regime when substituted for standard beef mince.

This project will provide preliminary evidence to support whether V2 plant-based mince could contribute to increased satiety following a meal, which may assist in a weight reduction dietary regime when substituted for standard beef mince.

The investigators specific hypotheses are:

H1: That participants will consume less KJ when consuming the V2 plant-based meal in comparison to the equivalent meal prepared with beef mince.

H2: That fullness will be maintained to the same extent following consumption of the V2 and meat-based meals, such that participants will not increase their consumption at the subsequent meal period to compensate for this energy deficit.

The null hypothesis is that a meal containing V2 plant-based meat is no more satiating than an equivalent meal containing beef mince.

This study is a single-blinded, randomised cross-over trial, designed to compare the effect of a meal prepared using V2 plant-based meat to an equivalent meal prepared with beef mince on the amount consumed in the current meal and objective and subjective measures of post-prandial satiety. The test meals will be formulated so that the meal will contain 45% of V2 plant-based meat or beef mince prior to the meal being cooked. Participants will be provided with a serving that is expected to be in excess of what they would be able to comfortably eat, and instructed to eat until comfortably full. The amount of the leftovers will be carefully weighed and used to calculate the volume, energy and macronutrient intake consumed.

180 mins after lunch (~3 pm), subjects will be presented with a standard cold buffet meal (including sliced bread, chicken, ham, cheese, mayonnaise, custard, yogurt, fruit salad and water) in excess of what they are expected to consume and allowed to eat ad libitum for up to 30 minutes. Participants will be asked to eat until they are comfortably full. The amount of each item consumed will be weighed and used to calculate total volume, energy and macronutrient intake.

ELIGIBILITY:
Inclusion Criteria:

1. Male individuals
2. Aged between ≥18 & ≤56 years at informed consent
3. Body mass index (BMI) ≥18.5 kg/m² and ≤27.5 kg/m² (confirmed during screening appointment)
4. Weight stable for last 6 months (< +/- 5kg change)*
5. Consume red meat regularly (at least 1 x week)
6. Willing to provide written Informed Consent
7. Be able to attend the CSIRO nutrition clinic for around 7 hours on two occasions across a two week period.

   * Self-reported

Exclusion Criteria:

1. Health conditions* that could affect appetite/food intake or require a prescribed diet such as gastrointestinal diseases [including, but not limited to diverticulitis, ulcerative colitis, Crohn's disease, or coeliac disease], type 1 or type 2 diabetes, cancer, renal or liver diseases
2. Gastrointestinal symptoms* (i.e. pain, reflux, diarrhea, or constipation), surgeries* (i.e. bariatric surgery such as gastric banding) or use of medications* (i.e. appetite suppressants, steroids) known to potentially affect energy intake, appetite, or gastrointestinal motor function
3. Known food allergies or intolerances to the study intervention products^
4. History of eating disorders*
5. Unable or unwilling to consume red meat
6. Current smoker (or history of smoking within the last six months)
7. History of or known presence of alcohol abuse or illicit drug use*
8. Received an investigational drug within 28 days prior to Visit 1 that in the opinion of the investigator may affect the applicant's ability to participate in the study or the study results *Self-reported, no clinical testing will be performed

Ages: 18 Years to 56 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Energy (kJ) consumed in test meals | 3 hours
  To determine whether a meal containing V2 plant-based meat is more satiating than an equivalent meal containing beef mince, as assessed by the energy (kJ) of the respective meals consumed to achieve fullness.
Visual Analogue Scale (VAS) | 4 hours
  Maintenance of satiety in the post-prandial period as measured by the VAS. Participants will indicate their perceived feelings of hunger, satiety, fullness and prospective food consumption at each time point on the VAS by moving the slider bar along a 10 mm line displayed on an iPad Question 1: How hungry do you feel? Answers to question 1: Please indicate how you are feeling at this moment by moving the slider bar to the appropriate point on each scale below (I am not hungry at all________________I have never been more hungry) Question 2: How satisfied do you feel? Answer to Q 2: I am completely empty_______________________________I cannot eat another bite.
  Question 3: How full do you feel? Anwer to Q3: Not at all full______________________Totally full Question 4: How much do you think you can eat? Answer to Q4: Nothing at all_________________________A lot.

SECONDARY OUTCOMES:
Energy consumed at subsequent buffet meal (kJ) | 4 hours
  measuring post-prandial satiety
Glucose (mmol/L) (plasma biomarker) | 4 hours
  measuring post-prandial satiety
insulin (pmol) (plasma biomarker) | 4 hours
  measuring post-prandial satiety
ghrelin (mcg) (plasma biomarker) | 4 hours
  measuring post-prandial satiety
cholecystokinin (CCK) (plasma biomarker) | 4 hours
  measuring post-prandial satiety
glucagon-like peptide-1 (GLP-1) (plasma biomarker) | 4 hours
  measuring post-prandial satiety

CONTACTS AND LOCATIONS:
Overall Officials: Bev Muhlhausler, BSc(Hons) PhD, Principal Investigator — Commonwealth Scientific and Industrial Research Organisation, Australia

IPD SHARING:
Plan to Share IPD: No